CLINICAL TRIAL: NCT01701453
Title: Smart Angioplasty Research Team: Safety of 6-month Duration of Dual Antiplatelet Therapy After Percutaneous Coronary Intervention in Patients With Acute Coronary Syndromes (SMART-DATE)
Brief Title: Safety of 6-month Duration of Dual Antiplatelet Therapy After Acute Coronary Syndromes (SMART-DATE)
Acronym: SMART-DATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-12-070
Record Dates: First submitted 2012-09-24; First posted 2012-10-05 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Acute Coronary Syndrome
Keywords: duration of DAPT
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 months group (Experimental): 6 months duration of P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel) treatment
  Interventions: Drug: P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel)
- 12 months or longer group (Experimental): 12 months or longer duration of P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel) treatment
  Interventions: Drug: P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel)

INTERVENTIONS:
Drug: P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel) — P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel)

SUMMARY:
1. Objective : To test the safety of 6 month-duration of dual antiplatelet therapy (DAPT) compared to conventional 12-month-or-longer duration after second-generation drug-eluting stent (DES) implantation in patients with acute coronary syndrome (ACS).
2. Hypothesis : A 6-month duration of DAPT is non-inferior to a conventional 12-month-or longer duration of DAPT at preventing the occurrence of major adverse cardiac and cerebrovascular events (MACCE) at 18-month after second-generation DES implantation in patients with ACS.

DETAILED DESCRIPTION:
1. Primary endpoint

   - MACCE, defined as a composite of all-cause mortality, myocardial infarction, and cerebrovascular events at 18 months after the index procedure.
2. Secondary endpoint

   * Individual components of the primary endpoint at 18-month after the index procedure
   * Definite/probable stent thrombosis, defined by the Academic Research Consortium (ARC) at 18-month after the index procedure.
   * Bleeding complication, defined by Bleeding Academic Research Consortium (BARC) type 2 to 5 at 18-month after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 20 years.
2. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving percutaneous coronary intervention and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
3. Subject must have a culprit lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation.
4. Subject must have clinical diagnosis of ACS that includes unstable angina and MI. The specific definitions of ACS, as follows; 1) ST-segment elevation MI (STEMI) : elevation of ST-segment more than 0.1 mV in 2 or more contiguous electrocardiographic (ECG) leads or new left bundle-branch block with elevated biomarkers of myocardial necrosis 2) Non-ST-segment elevation MI (NSTEMI) : Elevated biomarkers of myocardial necrosis (troponin or CK-MB > upper reference limit) with one of the following; (a) Transient ST-segment elevation or depression, or T-wave changes consistent with myocardial ischemia, (b) Identification of a culprit lesion at coronary angiography 3) Unstable angina : An accelerating pattern or recurrent episodes of chest pain at rest or with minimal effort and new ST-segment depression of at least 0.05 mV, or T wave inversion of at least 0.3 mV in at least 2 leads. The ECG criteria for unstable angina were based on the TACTICS-TIMI 18 trial.
5. Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥ 2.25 mm and ≤ 4.25 mm.
6. Target lesion(s) must be amenable for percutaneous coronary intervention

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Biolimus, Everolimus, Zotarolimus, and Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
2. Patients with active pathologic bleeding
3. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
4. Systemic (intravenous) Biolimus, everolimus, zotarolimus use within 12 months.
5. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
6. History of bleeding diathesis, known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
7. Noncardiac comorbid conditions are present with life expectancy <1 year or that may result in protocol noncompliance (per site investigator's medical judgment).
8. An elective surgical procedure is planned that would necessitate interruption of clopidogrel during the first 12 months post enrollment.
9. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2712 (Actual)
Dates: Start 2012-08; Primary Completion 2017-11 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
A composite of all-cause mortality, spontaneous myocardial infarction (MI), and cerebrovascular event | at 18-month after the index procedure
  defined as MACCE

SECONDARY OUTCOMES:
All-cause mortality | at 18-month after the index procedure
  Individual component of MACCE
Spontaneous MI | at 18-month after the index procedure
  Individual component of MACCE
Cerebrovascular event | at 18-month after the index procedure
  Individual component of MACCE
Stent thrombosis | at 18-month after the index procedure
  Definite or probable stent thrombosis defined by Academic Research Consortium (ARC)
Bleeding | at 18-month after the index procedure
  Bleeding Academic Research Consortium (BARC) type 2 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript

REFERENCES:
- [Derived] Song PS, Park YH, Oh JH, Song YB, Choi SH, Gwon HC, Cho DK, Rha SW, Bae JW, Jeong JO, Hahn JY; SMART-DATE and the SMART-CHOICE investigators. P2Y12 Inhibitor Monotherapy Versus Conventional Dual Antiplatelet Therapy or Aspirin Monotherapy in Acute Coronary Syndrome: A Pooled Analysis of the SMART-DATE and SMART-CHOICE Trials. Am J Cardiol. 2021 Jul 1;150:47-54. doi: 10.1016/j.amjcard.2021.03.053. Epub 2021 May 16. PMID 34011436
- [Derived] Kedhi E, Delewi R, Fabris E, De Luca G, Hermanides RS, van den Ent M, Buszman P, Zijlstra F, Song YB, Gwon HC, Hahn JY. Duration of dual antiplatelet therapy after myocardial infarction: Insights from a pooled database of the SMART-DATE and DAPT-STEMI trials. Atherosclerosis. 2020 Dec;315:55-61. doi: 10.1016/j.atherosclerosis.2020.11.003. Epub 2020 Nov 9. PMID 33227548
- [Derived] Choi KH, Song YB, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Oh JH, Cho DK, Lee JB, Doh JH, Kim SH, Jeong JO, Bae JH, Kim BO, Cho JH, Suh IW, Kim DI, Park HK, Park JS, Choi WG, Lee WS, Gwon HC, Hahn JY. Clinical Usefulness of PRECISE-DAPT Score for Predicting Bleeding Events in Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention: An Analysis From the SMART-DATE Randomized Trial. Circ Cardiovasc Interv. 2020 May;13(5):e008530. doi: 10.1161/CIRCINTERVENTIONS.119.008530. Epub 2020 May 1. PMID 32354228
- [Derived] Hahn JY, Song YB, Oh JH, Cho DK, Lee JB, Doh JH, Kim SH, Jeong JO, Bae JH, Kim BO, Cho JH, Suh IW, Kim DI, Park HK, Park JS, Choi WG, Lee WS, Kim J, Choi KH, Park TK, Lee JM, Yang JH, Choi JH, Choi SH, Gwon HC; SMART-DATE investigators. 6-month versus 12-month or longer dual antiplatelet therapy after percutaneous coronary intervention in patients with acute coronary syndrome (SMART-DATE): a randomised, open-label, non-inferiority trial. Lancet. 2018 Mar 31;391(10127):1274-1284. doi: 10.1016/S0140-6736(18)30493-8. Epub 2018 Mar 12. PMID 29544699